CLINICAL TRIAL: NCT04539340
Title: An Open-label Multi-cohort Dose-escalation Study to Evaluate the Tolerance, Safety, and Pharmacokinetics of GNR-055 (GENERIUM JSC, Russia) in Healthy Volunteers With a Single Intravenous Administration
Brief Title: A Multi-cohort Study of the Tolerance, Safety, and Pharmacokinetics of GNR-055 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDB-MPS-I
Record Dates: First submitted 2020-08-28; First posted 2020-09-07 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-08

CONDITIONS: Mucopolysaccharidosis Type II; Metabolic Diseases
Keywords: Mucopolysaccharidosis type II; Mucopolysaccharidoses; Metabolic Diseases; Lysosomal Storage Diseases; Carbohydrate Metabolism, Inborn; Metabolism, Inborn; Genetic Diseases, Inborn; Neurobehavioral Manifestations; Neurologic Manifestations; Genetic Diseases, X-Linked
MeSH Terms: conditions — Mucopolysaccharidosis II; Metabolic Diseases; Mucopolysaccharidoses; Lysosomal Storage Diseases; Genetic Diseases, Inborn; Neurobehavioral Manifestations; Neurologic Manifestations; Genetic Diseases, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 GNR-055 (0.3 mg/kg) (Other): GNR-055 (0.3 mg/kg) Single intravenous administration GNR-055
  Interventions: Biological: GNR-055
- Cohort 2 GNR-055 (0.5 mg/kg) (Other): GNR-055 (0.5 mg/kg) Single intravenous administration GNR-055
  Interventions: Biological: GNR-055
- Cohort 3 GNR-055 (1 mg/kg) (Other): GNR-055 (1 mg/kg) Single intravenous administration GNR-055
  Interventions: Biological: GNR-055
- Cohort 4 GNR-055 ( 2 mg/kg) (Other): GNR-055 ( 2 mg/kg) Single intravenous administration GNR-055
  Interventions: Biological: GNR-055
- Cohort 5 GNR-055 (3 mg/kg) (Other): GNR-055 (3 mg/kg) Single intravenous administration GNR-055
  Interventions: Biological: GNR-055

INTERVENTIONS:
Biological: GNR-055 — Single intravenous administration

SUMMARY:
It is a phase I open-label single-dose, dose-escalation cohort study to evaluate of the tolerance, safety, and pharmacokinetics of GNR-055 in healthy volunteers

DETAILED DESCRIPTION:
GNR-055 is intended for ERT in patient with Mucopolysaccharidosis type II (MPS II), or Hunter syndrome. MPS II is a lysosomal storage disease with an X-linked recessive inheritance type, which is characterized by a decrease in the activity of the lysosomal enzyme iduronate-2-sulfatase (I2S), caused by a mutation in the IDS gene. Enzyme deficiency leads to the accumulation of glycosaminoglycans (GAG) in lysosomes, mainly fractions of heparan and dermatan sulfates. Because of the insufficient activity of iduronate sulfatase participating in the first stage of catabolism of GAG, they accumulate in lysosomes of almost all types of cells of various tissues and organs. The disease is manifested by growth retardation, damage of many organs and systems, severe deformations of bones and joints, gross facial features, pathology of the respiratory and cardiovascular systems, damage to parenchymal organs (hepatosplenomegaly), and hearing impairment. A severe form of the disease occurs with the involvement of the nervous system in the pathological process, including mental retardation, behavior anomalies, and impaired motor function.

GNR 055 is a modified enzyme iduronate-2-sulfatase capable of penetrating the blood-brain barrier and thus it is expected to prevent neurodegenerative consequences and the development of cognitive deficit in the future that will allow achieving a significant improvement in the life quality and expectancy of patients with MPS II

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 50 years (inclusive) at the time of signing the Informed Consent Form;
* Body mass index (BMI) 18.5 to 30 kg/m2, body weight of 50 to 90 kg;
* A verified diagnosis as "healthy" (the diagnosis "healthy" is established on the basis of a detailed medical history, in the absence of deviations from normal values during a clinical examination, including measurement of blood pressure, respiratory rate, heart rate, body temperature, laboratory and instrumental (ECG) examination data);
* A written informed consent to participate in the study in accordance with applicable laws in place and compliance with all the procedures and requirements/restrictions provided for by the study protocol;
* Consent to use adequate methods of contraception (double barrier method-male or female (for partners of male research volunteers), condom with spermicide, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, cervical cap with spermicide).

Exclusion Criteria:

* Known hypersensitivity to idursulfase and/or to the medicinal product excipients;
* Burdened allergy history;
* Drug intolerance;
* History of seizures;
* Deposit injections or implants use of any other medicinal product three months before the Screening Visit;
* An unusual way of living (night working, extreme physical activity);
* Diarrhea dehydration, vomiting, or other causes within 24 hours before the Screening Visit;
* Deviations from the normal values of the clinical, laboratory, and ECG examinations;
* If there are acute or chronic diseases of the cardiovascular, bronchopulmonary, nervous, immune, and endocrine systems, diseases of the gastrointestinal tract, liver and biliary tract, kidney and urinary tract, blood and lymphatic system, a history of mental illness;
* Positive results for hepatitis B or C markers, human immunodeficiency virus (HIV), and syphilis;
* Acute infectious diseases less than four weeks before the Screening Visit;
* Regular administration of medicinal products less than two weeks before the Screening Visit;
* Systolic blood pressure (SBP) below 100 mm Hg or above 140 mm Hg; diastolic blood pressure (DBP) below 70 mm Hg or above 90 mm Hg; HR below 60 bpm or above 80 bpm;
* Blood donation (450 mL or more of blood or plasma) less than three months before the Screening Visit;
* Participation in human clinical studies of medicinal products less than three months before the Screening Visit;
* Consumption of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to 0.5 L of beer, 200 mL of dry wine, or 50 mL of strong spirits) OR history of alcoholism;
* Alcohol exhale positive test;
* Drug addiction, toxic substance abuse, a positive urine analysis for potent and narcotic substances, including cocaine, cannabis, amphetamine, barbiturates, benzodiazepines, and opioids;
* Smoking more than 10 cigarettes per day;
* Other reasons that, in the opinion of the investigator, prevent a volunteer from participating in the study or cause an unreasonable risk.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Day 7 ± 1
  Adverse events, Laboratory tests, Vital signs, Physical examination, 12-lead electrocardiogram, Allergic associated reaction, Infusion associated reaction, Antidrug antibody.

SECONDARY OUTCOMES:
Serum pharmacokinetic parameters of GNR-055 | Day 2
  Serum concentration GNR-055, Pharmacokinetic parameters
Cmax - Maximum Serum Concentration | Day 2
  Pharmacokinetic parameters
AUC - Area Under the Curve | Day 2
  Pharmacokinetic parameters
Т1/2 - Half-life | Day 2
  Pharmacokinetic parameters
Kel - Elimination rate constant | Day 2
  Pharmacokinetic parameters
MRT - Mean residence time | Day 2
  Pharmacokinetic parameters
Cl - Clearance | Day 2
  Pharmacokinetic parameters
Vz - volume of distribution | Day 2
  Pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Locations (1):
- FSAEI HE "I.M. Sechenov First Moscow State Medical University" of the Ministry of Health of Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No